CLINICAL TRIAL: NCT03165006
Title: CAMISS Retrospective Cohort - Effect of Interval Cancer and Screening Process on Survival and Disease-free Period in Breast Cancer
Brief Title: Effect of Interval Cancer and Screening Process on Survival and Disease-free Period in Breast Cancer
Status: Completed | Type: Observational
Sponsor: Parc de Salut Mar (Other)
Collaborators: Fondo de Investigacion Sanitaria (Other); European Regional Development Fund (Other); Red de Investigación en Servicios de Salud en Enfermedades Crónicas (Other)
Responsible Party: Principal Investigator, Maria Sala, MD, PhD, Parc de Salut Mar
Other Study IDs: CAMISS study
Record Dates: First submitted 2017-05-18; First posted 2017-05-24 (Actual); Last update posted 2017-05-24 (Actual); Status verified 2017-05

CONDITIONS: Breast Cancer
Keywords: Breast cancer, screening, survival
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Screened women with breast cancer
  Interventions: Procedure: Mode of detection: Cancer detected at screening; Procedure: Mode of detection: Interval cancer

INTERVENTIONS:
Procedure: Mode of detection: Cancer detected at screening — Cancers detected as a result of screening mammograms.
Procedure: Mode of detection: Interval cancer — Cancers diagnosed after a negative screening mammogram and before the next screening invitation (2 years in Spain)

SUMMARY:
This is a multicenter retrospective cohort of women participating in breast cancer screening programs in Spain between 2000 and 2009, with a cancer diagnosed during the screening or between the screening interval (interval cancer), specifically true interval cancers and false negatives. The investigators obtained woman-related information (including breast density), tumor-related information (including tumor phenotype), and follow-up information (including relapses, second neoplasms and vital status at the end of follow up (June 2014)). The objective is to evaluate the survival and disease-free period of women participating in screening programs for breast cancer with a cancer diagnosed during the screening or an interval cancer, specifically true interval cancers and false negatives.

This study is part of a broader project (CAMISS study), which also includes one prospective cohort (CAMISS Prospective cohort - Identifier in ClinicalTrials.gov: NCT02439554).

DETAILED DESCRIPTION:
The general objective for this study is to evaluate the survival and disease-free period of women participating in screening programs for breast cancer with a cancer diagnosed during the screening or an interval cancer, specifically true interval cancers and false negatives.

The cohort has information of women participating in breast cancer screening programs in Spain between 2000 and 2009, with a breast cancer diagnosed during the screening or between the screening interval (interval cancer), specifically true interval cancers and false negatives. The investigators obtained woman-related information (including breast density), tumor-related information (including tumor phenotype), and follow-up information (including relapses, second neoplasms and vital status at the end of follow up (June 2014)).

Expected results: Nowadays there are no results of cohort analysis of the diagnostic process of care that integrates all those different aspects. This study will complement the evaluation of population screening, specifically the interval cancer and the impact on survival and disease-free period taking into account relevant variables like breast density, tumor phenotype, clinical complications, readmissions, and the surgical approach.

This study is part of a broader project (CAMISS study) coordinated by the Evaluation of Health Services of Epidemiology and Public Health Group, which consists of two cohorts of women diagnosed with breast cancer: a prospective cohort (n=2,040 incident cases of breast cancer diagnosed in 18 hospitals of 5 Spanish regions) (Identifier in ClinicalTrials.gov: NCT02439554) and a retrospective cohort of screened women diagnosed with breast cancer between 2000 and 2009 in two Spanish regions (n=1,086).

The general objective of the CAMISS study is to evaluate different aspects of health care received by patients with breast cancer like the diagnostic process, treatment, complications, survival, costs and quality of life to provide information to improve the effectiveness and cost-effectiveness of interventions, reduce variability, have better predictive rules and increase the quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Women aged between 50 to 69 years with invasive or in situ breast cancer.

Exclusion Criteria:

* Women diagnosed with lobular carcinoma in situ.

Ages: 50 Years to 69 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Women participating at screening
Study Population: Women screened for breast cancer and diagnosed for breast cancer in the screening program (screen-detected cancer) or within the interval between 2 screening rounds (interval cancer)
Sampling Method: Non-Probability Sample
Enrollment: 1086 (Actual)
Dates: Start 2013-01-01 (Actual); Primary Completion 2014-06-30 (Actual); Study Completion 2015-12-31 (Actual)

PRIMARY OUTCOMES:
Mortality | From date of cancer diagnosis until the date of death from any cause, assessed up to 14 years
  Death from any cause

SECONDARY OUTCOMES:
Recurrences and second breast neoplasms | From date of cancer diagnosis until the date of the first recurrence or second breast neoplasm, whichever came first, assessed up to 14 years
Treatment-related complications | From the date of surgery until the end of follow-up, assessed up to 14 years.
Readmissions to hospital for reasons related to breast cancer | From the date of surgery until the end of follow-up, assessed up to 14 years.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Romero A, Tora-Rocamora I, Bare M, Barata T, Domingo L, Ferrer J, Tora N, Comas M, Merenciano C, Macia F, Castells X, Sala M; CAMISS Study Group. Prevalence of persistent pain after breast cancer treatment by detection mode among participants in population-based screening programs. BMC Cancer. 2016 Sep 15;16(1):735. doi: 10.1186/s12885-016-2768-1. PMID 27632982
- [Derived] Miret C, Domingo L, Louro J, Barata T, Bare M, Ferrer J, Carmona-Garcia MC, Castells X, Sala M. Factors associated with readmissions in women participating in screening programs and treated for breast cancer: a retrospective cohort study. BMC Health Serv Res. 2019 Dec 5;19(1):940. doi: 10.1186/s12913-019-4789-3. PMID 31805926
- See also: Related Info — http://www.camiss.info